CLINICAL TRIAL: NCT01062074
Title: Re-examination Study for General Vaccine Use to Assess the Safety Profile of GARDASIL in Usual Practice
Brief Title: GARDASIL Reexamination Study (V501-059)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: V501-059; 2010_005
Record Dates: First submitted 2010-02-02; First posted 2010-02-04 (Estimated); Results first posted 2014-03-27 (Estimated); Last update posted 2017-04-17 (Actual); Status verified 2017-03

CONDITIONS: Human Papillomavirus (HPV) Infection
MeSH Terms: conditions — Papillomavirus Infections; Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Korean Participants Vaccinated with GARDASIL: Females and males 9-26 years old who are vaccinated with GARDASIL in usual practice. The GARDASIL vaccination series consists of three 0.5-mL intramuscular injections. The second and third doses are to be administered 2 months and 6 months after the first dose, respectively.

SUMMARY:
This survey is conducted for preparing application materials for re-examination under the Pharmaceutical Affairs Laws and its Enforcement Regulation, its aim is to reconfirm the clinical usefulness of Gardasil through collecting the safety information according to the Re-examination Regulation for New Drugs.

ELIGIBILITY:
Inclusion Criteria:

* Females and males 9-26 years of age who Are Vaccinated With The First Dose Of Gardasil For The Prevention Of Any Disease Caused By Human Papillomavirus (e.g., Cervical Cancer, Genital Warts, etc.) Within Local Labeling

Exclusion Criteria:

* Participant Who Has A Contraindication To Gardasil According To The Local Label
* Participants Who Are Vaccinated With Gardasil Before Study Start

Ages: 9 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Females and males 9-26 Years Of Age who are vaccinated with GARDASIL in usual practice
Sampling Method: Probability Sample
Enrollment: 3605 (Actual)
Dates: Start 2007-09-28 (Actual); Primary Completion 2013-05-07 (Actual); Study Completion 2013-05-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=V501-059&kw=V501-059&tab=access

RESULTS

PARTICIPANT FLOW:
Groups:
- Korean Participants: Korean participants who received vaccination with GARDASIL, had Case Report Forms available, and did not violate the protocol
Period: Overall Study
Arm/Group | Korean Participants
Started | 3605
Completed | 3605
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Korean Participants
Number analyzed (Participants) | 3605
Age, Continuous [Mean (Standard Deviation); unit: Years] | 20.79 (4.02)
Age, Customized [Number; unit: Participants]
  <12 years | 122
  >=12 years and <19 years | 735
  >=19 years | 2748
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3549
  Male | 56

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Any Adverse Experience
Description: An adverse experience is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study vaccine, whether or not considered related to the use of the product. Any worsening of a preexisting condition which is temporally associated with the use of the study vaccine is also an adverse experience.
Time Frame: Up to 14 days after any GARDASIL vaccination
Population: Participants who received at least 1 vaccination with GARDASIL, had Case Report Forms available, and did not violate the protocol
Measure: Number; unit: Percent of participants
Arm/Group | Korean Participants
Number analyzed (Participants) | 3605
Percent of participants | 11.29

2. Primary Outcome: Percentage of Participants With Any Adverse Drug Reaction
Description: An adverse drug reaction was an adverse experience for which a causal relationship to the study drug could not be ruled out
Time Frame: Up to 14 days after any GARDASIL vaccination
Population: as for outcome 1
Measure: Number; unit: Percent of participants
Arm/Group | Korean Participants
Number analyzed (Participants) | 3605
Percent of participants | 9.02

ADVERSE EVENTS:
Time Frame: Up to 14 days after any GARDASIL vaccination
Arm/Group | Korean Participants
Serious Adverse Events (participants affected / at risk) | 0/3605
Other Adverse Events (participants affected / at risk) | 330/3605
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Korean Participants (N=3605)
Injection-site pain (General disorders) | 330 (504)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
With regard to surveillance results, any publication should be agreed by the sponsor in advance